CLINICAL TRIAL: NCT02477514
Title: A Multiple-Dose Study to Evaluate the Effects of Steady-State Tedizolid Phosphate Administration on the Pharmacokinetics and Safety of a Single Dose of Midazolam and Rosuvastatin
Brief Title: A Study to Evaluate the Effects of Tedizolid Phosphate on the Pharmacokinetics and Safety of Midazolam and Rosuvastatin (MK-1986-004)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1986-004; TR701-133 (Other: Cubist Protocol Number)
Record Dates: First submitted 2015-06-17; First posted 2015-06-22 (Estimated); Last update posted 2015-08-24 (Estimated); Status verified 2015-08

CONDITIONS: Skin Diseases, Bacterial
MeSH Terms: conditions — Skin Diseases, Bacterial | interventions — Midazolam; Rosuvastatin Calcium; tedizolid phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental Arm (Experimental): Day 1: participants will receive midazolam (2 mg); Day 3: participants will receive rosuvastatin (10 mg); Days 5-13: participants will receive tedizolid phosphate (200 mg); Day 14: participants will receive tedizolid phosphate (200 mg) plus midazolam (2 mg); Day 15: participants will receive tedizolid phosphate (200 mg); Day 16: participants will receive tedizolid phosphate (200 mg) plus rosuvastatin (10 mg); Day 17: participants will receive tedizolid phosphate (200 mg)
  Interventions: Drug: midazolam; Drug: rosuvastatin; Drug: tedizolid phosphate

INTERVENTIONS:
Drug: midazolam — 2 mg (1 mL of 2 mg/mL oral syrup) administered as a single dose on Days 1 and 14
Drug: rosuvastatin — 10 mg tablet administered as a single oral dose on Days 3 and 16
Drug: tedizolid phosphate — 200 mg oral tablet administered once daily on Days 5-17

SUMMARY:
The purpose of this study is to assess the effect of steady-state tedizolid phosphate on the single-dose pharmacokinetics of midazolam and rosuvastatin in healthy, adult participants.

ELIGIBILITY:
Inclusion Criteria:

* healthy, adult males or females (women of non-childbearing potential)
* continuous non-smokers who have not used nicotine-containing products for the previous 3 months

Exclusion Criteria:

* mentally or legally incapacitated or has significant emotional problems
* history or presence of clinically significant medical or psychiatric condition or disease
* history or presence of alcoholism or drug abuse within the past 2 years
* female participants who are pregnant, lactating, or of childbearing potential
* donated blood or had significant blood loss within 56 days prior to first dose of study drug
* plasma donation within 7 days prior to first dose of study drug

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2015-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Area under the concentration versus time curve, from 0 to last observed/measured non-zero concentration (AUC0-t) of midazolam alone or in combination with tedizolid phosphate | Days 1 and 14: pre-dose, 0.25, 0.5, 1, 1.5, 3, 4.5, 6, 8, 12, 24 hours
AUC0-t of rosuvastatin alone or in combination with tedizolid phosphate | Days 3 and 16: pre-dose, 1, 3, 4, 5, 6, 8, 16, 24, 36, 48 hours
Area under the concentration versus time curve from 0 to infinity (AUC0-inf) of midazolam alone or in combination with tedizolid phosphate | Days 1 and 14: pre-dose, 0.25, 0.5, 1, 1.5, 3, 4.5, 6, 8, 12, 24 hours
AUC0-inf of rosuvastatin alone or in combination with tedizolid phosphate | Days 3 and 16: pre-dose, 1, 3, 4, 5, 6, 8, 16, 24, 36, 48 hours
Maximum observed plasma concentration (Cmax) of midazolam alone or in combination with tedizolid phosphate | Days 1 and 14: pre-dose, 0.25, 0.5, 1, 1.5, 3, 4.5, 6, 8, 12, 24 hours
Cmax of rosuvastatin alone or in combination with tedizolid phosphate | Days 3 and 16: pre-dose, 1, 3, 4, 5, 6, 8, 16, 24, 36, 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC